CLINICAL TRIAL: NCT00860145
Title: Radiosurgery Versus Lobectomy for Temporal Lobe Epilepsy
Brief Title: Radiosurgery or Open Surgery for Epilepsy Trial
Acronym: ROSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: U01NS058634 (NIH); CRC; NINDS
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Epilepsy
Keywords: epilepsy; radiosurgery; temporal lobectomy
MeSH Terms: conditions — Epilepsy | interventions — Radiosurgery; Anterior Temporal Lobectomy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- radiosurgery (Experimental): Radiosurgical treatment of the medial temporal lobe
  Interventions: Procedure: radiosurgery
- temporal lobectomy (Active Comparator): Resection of medial temporal lobe
  Interventions: Procedure: temporal lobectomy

INTERVENTIONS:
Procedure: radiosurgery — The stereotaxic frame will be secured to the skull with four pins. Patients will be taken to the MRI unit and receive a stereotaxic MRI. MRI data will be transferred to the Gamma Knife computer. Each patient will receive radiation to the mesial temporal lobe during a single treatment session. The amygdala and anterior 2cm of the hippocampus as well as the immediately adjacent parahippocampal gyrus will be included in the radiosurgical target. Patients will receive 24Gy to the 50% isodose line using an unlimited number of isocenters. The brainstem and optic nerve plus chiasm will receive less than 10 Gy and 8 Gy, respectively. After treatment, the stereotaxic frame will be removed from the patient's head.
  Other Names: Gamma Knife
  Arms: radiosurgery
Procedure: temporal lobectomy — The temporal lobectomy will be performed under general anesthesia. The superior temporal gyrus will be resected to a minimal degree (typically between 1 and 2cm) and the middle and inferior temporal gyri will be resected to approximately 3cm.The minimum amount of lateral temporal cortex required to perform an aggressive resection of medial temporal structures will be performed. The temporal portion of the amygdala and the anterior two to three cm of the hippocampus will be resected. In addition, nearby entorhinal cortex will be removed.
  Arms: temporal lobectomy

SUMMARY:
This study will compare radiosurgery (focused radiation, Gamma Knife Radiosurgery) with temporal lobectomy (standard surgical care) as a treatment of temporal lobe epilepsy. Patients who have seizures that begin in their temporal lobe that are not controlled with medications into the trial will be offered entry. Patients with a high likelihood of having their seizures controlled with open surgery will have treatment randomized between the standard surgery and radiosurgery. A prior study has shown that focused radiation (radiosurgery) may also reduce or eliminate seizures arising from the temporal lobe. The main study hypothesis is that radiosurgery is as safe and effective as temporal lobectomy in treating patients with seizures arising from the medial temporal lobe.

DETAILED DESCRIPTION:
The purpose of this study is to compare the effectiveness of Gamma Knife radiosurgery with temporal lobectomy in the treatment of patients with drug resistant temporal lobe epilepsy. Aim 1 is designed to compare the seizure-free outcomes and morbidity of radiosurgery for patients with drug resistant temporal lobe epilepsy with those of open temporal lobectomy. Our primary hypothesis is that radiosurgery will be non-inferior to lobectomy with respect to seizure-free rates at 25-36 months following therapy (one-year of seizure freedom beginning 2 years after treatment).

Aim 2 is designed to compare the neuropsychological outcomes in patients undergoing radiosurgery and temporal lobe surgery, in particular with respect to verbal memory function for language-dominant hemisphere treated patients. Our hypothesis is that patients treated for speech-dominant temporal lobe seizures with temporal lobectomy will show greater reduction in verbal memory than patients treated with radiosurgery.

Aim 3 is designed to determine what changes occur in the quality of life of patients with temporal lobe epilepsy following radiosurgical treatment as compared with open surgery. Our primary hypothesis is that there will be improvements (comparing baseline with 3 years post-treatment) in quality of life measures in both groups. Our secondary hypothesis is that both open surgery and radiosurgery subjects will undergo transient reductions in quality of life measures caused by treatment effects during the first year following treatment, but that quality of life will improve for subjects who become seizure-free, independent of treatment group.

Aim 4 is designed to compare the cost-effectiveness of radiosurgery compared with open surgery. Specifically, the marginal cost-utility ratio will fall below $50,000/QALY, a threshold thought to indicate that outcomes are considered worth the cost.

ELIGIBILITY:
Inclusion and Exclusion Criteria:

Adults (18 years and older) of either gender who would otherwise be eligible for temporal lobe resection will be offered enrollment for randomization to RS or ATL.

1. Seizure type: Patients must have simple and/or complex partial seizures with or without secondary generalization.
2. Seizure Frequency: Patients must have at least 3 complex partial seizures during the 3 month (12 week) baseline seizure diary period with at least 1 of 3 seizures occurring within the last 2 months (8 weeks).
3. Patients with electrographic evidence of seizures arising from one temporal lobe, with radiographic evidence of mesial temporal sclerosis in the same temporal lobe will be included. Patients with normal MRIs, bilateral hippocampal damage, or cortical lesion will be excluded.
4. Subjects should be on stable doses of antiepileptic medications for at least 3 months prior to treatment.
5. All female patients of childbearing age will have documented that they are using a safe and effective means of birth control and will have a negative urine pregnancy test completed within 1 week prior to their treatment.
6. Patients should be able to understand the potential benefits and risks of this therapy and be able to understand the protocol and sign their own consent forms. For these reasons, only patients 18 years and older and with I.Q. greater than or equal to 70 will be included.
7. Patients with any focal neurologic deficit that would make it difficult to detect a new radiation-associated injury will be excluded. All patients will receive formal visual field testing (Humphrey) and patients with visual field deficits will be excluded.
8. Patients with radiographic evidence of other pathologies such as vascular malformations or tumors will be excluded.
9. Patients with diabetes mellitus or hypertension will be excluded from this study because radiation injury to the brain is more common in these patients.
10. Subjects should not have significant psychiatric conditions that would make accurate assessment of seizure frequency difficult, as judged by the principal investigator. Such conditions include a history of non-epileptic seizures, psychosis (other than post-ictal psychosis) and severe mood disorders including suicide attempt within past 12 months or noncompliance with psychotropic medications.
11. Patients with a history of significant past or present medical disorders determined severe enough to prevent participation in a surgical trial by the principal investigator are excluded.
12. Patients with any progressive neurological disorder (such as multiple sclerosis or systemic lupus erythematosis) are excluded.
13. Patients with a history of poor compliance with past antiepileptic drug therapy as judged by the principal investigator are excluded.
14. Patients with a recent history of abusing drugs or alcohol with significance as judged by the principal investigator are excluded.
15. Patients who are receiving any investigational drugs at the time of enrollment are excluded.
16. Patients with current use of vigabatrin are excluded. Past use does not exclude a patient pending a normal formal visual field test.
17. Patients with currently functioning vagal nerve stimulators (VNS) are excluded. Past use does not exclude a patient as long as the device is explanted. Indwelling VNS electrodes are permitted in agreement with each center's policies on brain MRI imaging.
18. Patients who can not be anticipated to participate for the full 36 months of the trial will be excluded.
19. Native English speakers from the U.S. or other English speaking countries or patients who learned English before age 5 and were educated in English. Spanish speaking patients can be included as long as the study site can provide an officially translated (IRB approved) consent form in Spanish. Non-Spanish speaking patients with English as a second language (ESL) and/or non-English and non-Spanish speaking patients can be included only under the following conditions: 1) the study site must be able to have the consent form translated into the patient's native language using an official translator, and 2) the study site's neuropsychologist must be willing and able to assess the patient at baseline and post-treatment at 12, 24, and 36 months in that patient's native language to ensure the patient's safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2009-09; Primary Completion 2016-06-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is freedom from seizures. The primary goal of Specific Aim 1 is to demonstrate that the 3-year seizure-free rate of radiosurgery is not inferior to that of temporal lobectomy between 24 and 36 months following treatment. | 3 years

SECONDARY OUTCOMES:
Specific Aim 2 is designed to show that patients treated for speech-dominant temporal lobe seizures with temporal lobectomy will show greater reduction in verbal memory than patients treated with radiosurgery. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Ver Hoef, MD, Principal Investigator — University of Alabama at Birmingham; Guy McKhann, MD, Principal Investigator — Columbia University; Vincenta Salanova, MD, Principal Investigator — Indiana University; Thomas Pittman, MD, Principal Investigator — University of Kentucky; Andriana E. Palade, MD, Principal Investigator — West Virginia University; Aviva Abosch, MD, PhD, Principal Investigator — University of Minnesota; Anto Bagic, MD, MSc, Principal Investigator — University of Pittsburgh, Medical School; Robert L Beach, MD, PhD, Principal Investigator — Upstate Medical University; Evelyn S Tecoma, MD, PhD, Principal Investigator — University of California, San Diego; Christi N Heck, MD, PhD, Principal Investigator — University of Southern California; John W Miller, MD, PhD, Principal Investigator — University of Washington; Nathan B Fountain, MD, Principal Investigator — University of Virginia; Paul Garcia, MD, Principal Investigator — University of California, San Francisco; Nicholas M. Barbaro, MD, Principal Investigator — University of California, San Francisco; Mark S Quigg, MD, MSc, Principal Investigator — University of Virginia; Kenneth D Laxer, MD, Study Chair — California Pacific Medical Center; John Langfitt, MA, PhD, Study Chair — University of Rochester; Penny Sneed, MD, Study Chair — University of California, San Francisco; Michael W McDermott, MD, Study Chair — University of California, San Francisco
Locations (14):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Indiana University, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University, New York, New York
  - State University of New York, Upstate Medical Center, Syracuse, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - University of Washington, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
- All India Institute of Medical Sciences (AIIMS), New Delhi, India

IPD SHARING:
Plan to Share IPD: Yes
Preliminary report 12/2016 at the American Epilepsy Society meeting. Full paper to follow.

REFERENCES:
- [Background] Barbaro NM, Quigg M, Broshek DK, Ward MM, Lamborn KR, Laxer KD, Larson DA, Dillon W, Verhey L, Garcia P, Steiner L, Heck C, Kondziolka D, Beach R, Olivero W, Witt TC, Salanova V, Goodman R. A multicenter, prospective pilot study of gamma knife radiosurgery for mesial temporal lobe epilepsy: seizure response, adverse events, and verbal memory. Ann Neurol. 2009 Feb;65(2):167-75. doi: 10.1002/ana.21558. PMID 19243009